CLINICAL TRIAL: NCT00879554
Title: A Multicenter, Open-Label, 2-Stage, Phase 1, Clinical Safety, Pharmacokinetic, And Pharmacodynamic Study Of CVX-045, A Thrombospondin-1 Mimetic, Anti-Angiogenic Agent, In Patients With Advanced Solid Tumors
Brief Title: A Safety And Pharmacokinetic Study With CVX-045 In Patients With Advanced Solid Tumors
Acronym: CVX-045-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1121003
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Advanced Solid Tumors; Neoplasms; Carcinoma; Cancer; Malignancy
Keywords: Phase 1; Solid Tumors; CVX-045
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: CVX-045

INTERVENTIONS:
Biological: CVX-045 — Weekly, intravenous dose

SUMMARY:
The purpose of the study is to determine safety and tolerability of CVX-045 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced solid tumors unresponsive to currently available therapies, or for which there is no standard therapy.
* Adequate coagulation, liver and renal function.
* Candidate for DCE-MRI evaluation.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1.

Exclusion Criteria:

* Evidence of bleeding problems.
* Uncontrolled hypertension.
* Certain gastrointestinal problems including fistula and abscess.
* Patients with primary brain cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine safety and tolerability of CVX-045 as weekly intravenous (IV) infusions in adult patients with advanced solid tumors | Throughout duration of study
To identify and characterize CVX-045-related adverse events (AEs) | Throughout duration of study

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics (PK) of CVX-045 | Days 1, 4, 8, 15, 29
To determine a recommended Phase 2 dose of CVX-045 | End of study
To evaluate the potential for immunogenicity of CVX-045 | Days 1, 15, 1st day of every subsequent cycle, EOS, 30 Day FU
To document any preliminary evidence of antitumor activity | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1121003&StudyName=A%20%20Safety%20And%20Pharmacokinetic%20Study%20With%20CVX-045%20In%20Patients%20With%20Advanced%20Solid%20Tumors